CLINICAL TRIAL: NCT03317665
Title: Prospective, Observational Trial of Biological or Prosthetic Mesh for Open Ventral Hernia Repair
Brief Title: Observational Biologic or Prosthetic Mesh
Status: Terminated | Type: Observational
Why Stopped: Premature termination due to cease of funding
Sponsor: University of South Florida (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: CA2017-003
Record Dates: First submitted 2017-10-10; First posted 2017-10-23 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Ventral Incisional Hernia
Keywords: biologic; prosthetic; mesh
MeSH Terms: interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard of care: Mesh for hernia repair: Standard of care products used by the Investigator for open ventral hernia repair procedure
  Interventions: Device: Mesh for hernia repair

INTERVENTIONS:
Device: Mesh for hernia repair — Permacol, Parietex, Progrip, Strattice Perforated, and Surgimend.

SUMMARY:
The purpose of this study is to assess the incidence of hernia recurrence with the use of biologic and prosthetic mesh in ventral hernia repair.

DETAILED DESCRIPTION:
Incisional hernias are very common, leading to over 380,000 operative repairs done annually. Despite the commonality of this problem, there has been no single operative repair that has become the standard. This is due to the high recurrence rates with all types of repairs, especially primary suture repair. Because of this, most repairs are done with some type of mesh, either made out of a prosthetic material or biologic material. Mesh repairs, however, have their own problems, namely surgical site infections and potential bowel erosion. Potential complications associated with prosthetic mesh for hernia repairs include: adverse reactions to the mesh, mesh erosion, stricture formation, adhesions resulting in bowel obstruction, enterocutaneous fistulas, injuries to nearby organs, nerves or blood vessels, infection, chronic pain and hernia recurrence. Potential complications associated with biological mesh include: adverse inflammatory response, laxity, eventration, and recurrent herniation. To address these mesh related complications, the separation of components technique was developed to reduce tension on the midline repair and the underlay technique was developed to place the mesh in the retrorectus space. Nevertheless, this technique still has a significant recurrence rate.

Therefore, the purpose of this study is to evaluate the effectiveness of biological or prosthetic mesh in incisional hernia repair, by assessing the associated rates of hernia recurrence and complications.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients > 21 years old.
* Able to provide informed consent in English or Spanish.
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study, if applicable.
* Allergy or hypersensitivity to materials in porcine-based study products, prosthetic or biological meshes, or personal preference.
* Male and female patients ≤ 21 years old
* History of drug addiction (recreational drugs, prescription drugs or alcohol) that in the Investigator's opinion may interfere with protocol assessments and/or the subject's ability to complete the required follow up.
* Serious or active medical or psychiatric condition which, in the opinion of the Investigator, may interfere with treatment, assessment, or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring open ventral hernia repair.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of ventral hernia recurrence | 2 years from study ventral hernia repair

SECONDARY OUTCOMES:
Time to ventral hernia recurrence | 2 years from study ventral hernia repair
Incidence of wound complications | 90 days from study ventral hernia repair
  Complications of interest: surgical site infections, seroma formation, and wound dehiscence or skin separation
Incidence of enterocutaneous fistula formation | 2 years from study ventral hernia repair
Mean Carolinas Comfort Scale score | 2 years from study ventral hernia repair
  Patient-centered outcome assessing hernia symptoms - minimum score 0 and maximum total score 115
Mean Visual Analog Scale score | 2 years from study ventral hernia repair
  Patient-centered outcome - pain score measured by a line in millimeters (0 for no pain and 10 for worst pain imaginable)
Mean mesh deployment time | during surgery
  Defined as the time mesh preparation starts to time mesh placement ends
Mean procedure time | during surgery
  Defined as time of incision to time of closure
Mean total cost of hospitalization for primary admission | From date of surgery to date of hospital discharge (approximately 3 days)
  Defined as cost from surgery to hospital discharge
Mean total cost of surgery for primary admission | during surgery
  Defined as cost from preoperative preparation to anesthesia discharge
Mean total cost of narcotic usage for primary admission | From date of surgery to date of hospital discharge (approximately 3 days)
  Defined as cost from narcotic use from surgery to hospital discharge
Mean total cost of readmissions | 2 years from study ventral hernia repair
  any hospital readmissions related to ventral hernia complications or recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Vic Velanovich, MD, Principal Investigator — University of South Florida
Locations (3):
- United States (3):
  - Tampa General Hospital, Tampa, Florida
  - University of South Florida - South Tampa Campus, Tampa, Florida
  - University of South Florida Morsani Center for Advanced Health Care, Tampa, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fekkes JF, Velanovich V. Amelioration of the effects of obesity on short-term postoperative complications of laparoscopic and open ventral hernia repair. Surg Laparosc Endosc Percutan Tech. 2015 Apr;25(2):151-7. doi: 10.1097/SLE.0000000000000100. PMID 25222715
- [Background] Poulose BK, Shelton J, Phillips S, Moore D, Nealon W, Penson D, Beck W, Holzman MD. Epidemiology and cost of ventral hernia repair: making the case for hernia research. Hernia. 2012 Apr;16(2):179-83. doi: 10.1007/s10029-011-0879-9. Epub 2011 Sep 9. PMID 21904861
- [Background] Fischer JP, Wink JD, Tuggle CT, Nelson JA, Kovach SJ. Wound risk assessment in ventral hernia repair: generation and internal validation of a risk stratification system using the ACS-NSQIP. Hernia. 2015 Feb;19(1):103-11. doi: 10.1007/s10029-014-1318-5. Epub 2014 Dec 4. PMID 25472771
- [Background] Zhou XH, Melfi CA, Hui SL. Methods for comparison of cost data. Ann Intern Med. 1997 Oct 15;127(8 Pt 2):752-6. doi: 10.7326/0003-4819-127-8_part_2-199710151-00063. PMID 9382393
- [Result] Holihan JL, Alawadi Z, Martindale RG, Roth JS, Wray CJ, Ko TC, Kao LS, Liang MK. Adverse Events after Ventral Hernia Repair: The Vicious Cycle of Complications. J Am Coll Surg. 2015 Aug;221(2):478-85. doi: 10.1016/j.jamcollsurg.2015.04.026. Epub 2015 May 9. PMID 26206646
- [Result] Heniford BT, Walters AL, Lincourt AE, Novitsky YW, Hope WW, Kercher KW. Comparison of generic versus specific quality-of-life scales for mesh hernia repairs. J Am Coll Surg. 2008 Apr;206(4):638-44. doi: 10.1016/j.jamcollsurg.2007.11.025. Epub 2008 Feb 1. PMID 18387468
- [Result] Nielsen K, Poelman MM, den Bakker FM, van der Ploeg T, Bonjer HJ, Schreurs WH. Comparison of the Dutch and English versions of the Carolinas Comfort Scale: a specific quality-of-life questionnaire for abdominal hernia repairs with mesh. Hernia. 2014 Aug;18(4):459-64. doi: 10.1007/s10029-013-1173-9. Epub 2013 Oct 29. PMID 24166693
- [Result] FitzGerald JF, Kumar AS. Biologic versus Synthetic Mesh Reinforcement: What are the Pros and Cons? Clin Colon Rectal Surg. 2014 Dec;27(4):140-8. doi: 10.1055/s-0034-1394155. PMID 26106284
- [Result] Aravot DJ, Banner NR, Khaghani A, Fitzgerald M, Radley-Smith R, Mitchell AG, Yacoub MH. Cardiac transplantation in the seventh decade of life. Am J Cardiol. 1989 Jan 1;63(1):90-3. doi: 10.1016/0002-9149(89)91082-5. PMID 2642367